CLINICAL TRIAL: NCT00287105
Title: An Open-label, Phase II Study to Explore the Safety and Efficacy of Imatinib With Chemotherapy in Pediatric Patients With Ph+ / BCR-ABL+ Acute Lymphoblastic Leukemia (Ph+ALL)
Brief Title: Safety and Efficacy of Imatinib Added to Chemotherapy in Treatment of Ph+ Acute Lymphoblastic Leukemia in Children
Acronym: ESPHALL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Collaborators: Ministry of Health, France (Other Government); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EUDRACT 2004-001647-30; PHRC/04-04; CIC0203/043
Record Dates: First submitted 2006-02-03; First posted 2006-02-06 (Estimated); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Acute Lymphoblastic Leukemia; Philadelphia Chromosome
Keywords: Chemotherapy; Leukemia; Children; Philadelphia chromosome; Protein-tyrosine kinase inhibitor
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Philadelphia Chromosome; Leukemia | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Good risk Ph+ALL (Other): For protocols which adopt a steroid prephase: patients who are Prednisone-good responder and achieve CR after the induction course. For protocols which do not adopt steroid prephase: patients who have M1/M2 BM at day 15 or M1 BM at day 21 and achieve CR after the induction course. Expected stratification in this group: 70-75%.
  Interventions: Drug: Standard chemotherapy + Imatinib
- Poor risk Ph+ALL (Other): For protocols which adopt a steroid prephase: patients who are Prednisone poor-responders. For protocol which do not adopt a steroid prephase: patients who have M3 BM at day 15 or M2/M3 BM at day 21. For all protocols: patients who do not achieve CR after the induction course. Expected stratification: 25-30%.
  Interventions: Drug: Standard chemotherapy + Imatinib

INTERVENTIONS:
Drug: Standard chemotherapy + Imatinib — Patients receive Imatinib together with the standard chemotherapy regimen of phase IB and after each of three consecutive blocks of the standard chemotherapy in the consolidation phase
  Other Names: Glivec; Gleevec

SUMMARY:
The purpose of this study is to determine whether Imatinib is safe and effective in association with intensive treatment of Ph+ALL in children.

DETAILED DESCRIPTION:
Recent advances in treatment have increased the cure of childhood ALL to 75% or better. However, attempts to improve results for resistant subtypes of ALL, such as Ph+ ALL, have been largely unsuccessful. Imatinib, an inhibitor of protein-tyrosine kinases, is currently being tested in several phase I, II and III trials covering most Chronic Myeloid Leukemia patient populations and patients with overtly relapsed or refractory Ph+ALL. Pediatric patients with Ph+ALL will receive Imatinib, added to intensive, post-induction BFM-type chemotherapy. The endpoint will be the evaluation on the long-term clinical outcome, in particular on the Disease Free Survival (DFS).

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents aged 1 to 17 years at diagnostic
* Documented Ph+ ALL
* Eligibility for the current local prospective therapeutic study of childhood ALL
* Informed consent given by the parents or by legal guardian

Exclusion Criteria:

* Abnormal hepatic functions
* Abnormal renal functions
* Active systemic bacterial, fungal or viral infection

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 49 (Actual)
Dates: Start 2005-12 (Actual); Primary Completion 2016-03-30 (Actual); Study Completion 2017-03-03 (Actual)

PRIMARY OUTCOMES:
Disease free survival (DFS). DFS will be calculated as the time from inclusion to either one of the following events: relapse, death in CCR, second malignancies. | 2 years

SECONDARY OUTCOMES:
Compare long term outcome between patients treated by BFM-chemotherapy and patient undergoing more intensive chemotherapy (protocole COGAALL0031 : Children Oncology Group-USA). | 2 years
Long-term clinical outcome : Disease free survival (DFS), Event-Free Survival (EFS) and Overall Survival (OS) in each risk groups. | 2 years
Pattern of molecular response (MRD) | 5 time points between S4 and S22
Conversion rate to CR in patients resistant to the first part of the induction phase of chemotherapy included in the Poor-risk group. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Biondi, MD, Study Director — Ospedale S. Gerardo - Monza; Virginie Gandemer, MD, Principal Investigator — Rennes University Hospital
Locations (22):
- France (22):
  - Service d'hématologie pédiatrique CHRU, Amiens
  - Service hématologie pédiatrique Hôpital Saint-Jacques, Besançon
  - Service d'hémato-oncologie - Hôpital des Enfants Pellegrin, Bordeaux
  - Hôpital Morvan, Brest
  - Hématologie oncologie pédiatrique-CHU Caen, Caen
  - Hémato-Oncologie et Thérapie Cellulaire Pédiatrique - Hôtel Dieu, Clermont-Ferrand
  - Hémato-Oncologie Pédiatrique - Hôpital d'Enfants, Dijon
  - Pédiatrie CHU - Hôpital Nord, Grenoble
  - Hôpital Jeanne de Flandre, Lille
  - Limoges University Hospital, Limoges
  - Hôpital DEBROUSSE Institut d'hématologie et d'oncologie pédiatrique, Lyon
  - Hôpital Arnaud de Villeneuve, Montpellier
  - Hématologie Pédiatrique - Hôpital Trousseau, Paris
  - Hémato-immunologie-Robert Debré, Paris
  - Hématologie Hôpital Jean Bernard, Poitiers
  - Hématologie pédiatrique-Hopital américain, Reims
  - Service d'hématologie pédiatrique - Hôpital Sud, Rennes
  - Service d'Immuno Hémato Oncologie Pédiatrique - Hôpital Charles Nicolle, Rouen
  - Hématologie, Oncologie pédiatrique-CHU Saint Etienne, Saint-Etienne
  - Hopital des enfants, Toulouse
  - CHU- Centre Gatien de Clocheville, Tours
  - Hôpital d'enfants, Vandœuvre-lès-Nancy

REFERENCES:
- [Result] Biondi A, Schrappe M, De Lorenzo P, Castor A, Lucchini G, Gandemer V, Pieters R, Stary J, Escherich G, Campbell M, Li CK, Vora A, Arico M, Rottgers S, Saha V, Valsecchi MG. Imatinib after induction for treatment of children and adolescents with Philadelphia-chromosome-positive acute lymphoblastic leukaemia (EsPhALL): a randomised, open-label, intergroup study. Lancet Oncol. 2012 Sep;13(9):936-45. doi: 10.1016/S1470-2045(12)70377-7. Epub 2012 Aug 14. PMID 22898679
- [Result] Biondi A, Gandemer V, De Lorenzo P, Cario G, Campbell M, Castor A, Pieters R, Baruchel A, Vora A, Leoni V, Stary J, Escherich G, Li CK, Cazzaniga G, Cave H, Bradtke J, Conter V, Saha V, Schrappe M, Grazia Valsecchi M. Imatinib treatment of paediatric Philadelphia chromosome-positive acute lymphoblastic leukaemia (EsPhALL2010): a prospective, intergroup, open-label, single-arm clinical trial. Lancet Haematol. 2018 Dec;5(12):e641-e652. doi: 10.1016/S2352-3026(18)30173-X. PMID 30501871
- [Derived] Tasian SK, Peters C. Targeted therapy or transplantation for paediatric ABL-class Ph-like acute lymphocytic leukaemia? Lancet Haematol. 2020 Dec;7(12):e858-e859. doi: 10.1016/S2352-3026(20)30369-0. No abstract available. PMID 33242441
- See also: Primary Publication — https://pubmed.ncbi.nlm.nih.gov/30501871/